26.02.2025

Title: Methyl Alcohol Intoxication as a Public Health Issue: A 3-Year Retrospective Analysis

Yeliz Bilir\*, Banu Çevik\*, Akın Bilir\*, Elif Bombacı\*.

\*Department of Intensive Care, Kartal Dr Lütfi Kırdar City Hospital, İstanbul, Turkey

\*Corresponding author: Yeliz Bilir, M.D.

E-mail: dryelizbilir@yahoo.com

Address: Kartal Dr. Lütfi Kırdar City Hospital, D-100 Güney Yanyol No:47 Cevizli Mevkii

34865 Kartal / İSTANBUL

Phone: +90 5326657976

**Number of Tables: 5** 

**Number of Figures: 2** 

Word count: 2500

NCT Number: Not Available

Keywords: Methanol, Intoxication, Treatment, Outcomes.

## **Statistical Analysis:**

Statistical analyses were conducted using SPSS 27.0.1 (IBM, Armonk, NY, USA). Continuous variables were presented as mean  $\pm$  standard deviation (SD), while categorical variables were expressed as frequency (n) and percentage (%). The normality of continuous data was assessed via the Shapiro-Wilk and Kolmogorov-Smirnov tests, histograms, and skewness-kurtosis values. Student's t-test and Mann-Whitney U test were used for parametric and nonparametric comparisons, respectively. Categorical variables were analyzed using Pearson's chi-square test or Fisher's exact test (for n < 5). Independent risk factors for mortality were identified using the area under the curve (AUC) and ROC analysis to determine optimal mortality predictors. Odds ratios (OR) with 95% confidence intervals (CI) were calculated, and statistical significance was set at p  $\leq$  0.05.